CLINICAL TRIAL: NCT04672044
Title: Feasibility of Combination Exercise and Neuromodulation Rehabilitation to Improve Post-stroke Chronic Pain
Brief Title: TMS and Exercise for Post-stroke Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B3612-P; I21RX003612 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Chronic Post-stroke Headache
Keywords: Vascular Headaches; post-stroke headache
MeSH Terms: conditions — Vascular Headaches | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: Feasibility of a double-blind sham-controlled intervention
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- active rTMS+Exercise (Active Comparator): active rTMS
  Interventions: Device: Active rTMS and exercise
- sham rTMS+Exercise (Sham Comparator): sham rTMS
  Interventions: Combination Product: Sham rTMS+Exercise

INTERVENTIONS:
Device: Active rTMS and exercise — active
  Arms: active rTMS+Exercise
Combination Product: Sham rTMS+Exercise — sham
  Arms: sham rTMS+Exercise

SUMMARY:
There are over 7 million people living with stroke in the United States. Per year, approximately 17,000 Veterans are admitted to the VA for acute stroke. Chronic pain after stroke can occur between 10-50% of stroke survivors. Post-stroke pain (PSP) can lead to further complications in a stroke survivor's recovery. Exercise has improved PSP and associated symptoms such as mobility, fatigue, and quality of life. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive technique using electromagnetic induction for cortical neurostimulation. The use of rTMS has been explored shown to be effective in treating chronic PSP but is limited in effect duration. Our proposal will test the hypothesis that rTMS is feasible and safe to be paired with exercise. Additionally, the investigators believe a complementary effect can develop to enhance the neurostimulation duration of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veteran of US military 19 years of age
* Signed informed consent
* Minimum of 3-months since time of stroke and medically stable
* Headache has persisted for >3 months after stabilization of the stroke
* Ability to walk or tolerate recumbent cycle ergometry for 10 mins without assistance
* Stable pain medication regimen for 1 month prior to study
* Females of child-bearing potential (i.e. not postmenopausal or surgically sterile) must be using a medically acceptable method of birth control and should not be pregnant nor have plans for pregnancy or breastfeeding during the study
* Completed diagnostic, maximal graded exercise test including 12-lead ECG and indirect calorimetry (i.e. oxygen uptake, minute ventilation, respiratory exchange ratio, etc.)
* Minimum pain intensity of 30 on the Mechanical Visual Analogue Scale on average with pain symptoms.

Exclusion Criteria:

* Moderate to severe cognitive impairment (Montreal Cognitive Assessment score <16/30)
* Pre-stroke modified Rankin >2
* History of seizures
* Presence of any standard TMS or MRI contraindications (see human subjects)
* Current diagnosis of DSM-5-defined bipolar disorder I, schizophrenia, schizoaffective disorder, or obsessive-compulsive disorder
* Diagnosis of moderate or severe substance use disorder (except for caffeine and nicotine) during the preceding 3 months (Participants must agree to abstain from illicit drugs during the study)
* Increased risk of suicide that necessitates inpatient treatment or warrants additional therapy excluded by the protocol; and/or intensity of suicidal ideation (Type 4 or Type 5) or any suicidal behavior in the past 3 months on Columbia Suicide Severity Rating Scale (C-SSRS)
* Litigating for compensation for a psychiatric disorder

  * Veterans who are in the process of applying for or receiving VA service-connected disability are eligible
* Current enrollment in another intervention trial for pain or stroke
* Persons imprisoned, of minor age, diagnosed with terminal illness, or require surrogate for consent
* Fails baseline exercise screening activities
* Persistent post-stroke headaches not better accounted for by another diagnosis
* Is unable to reliably attend intervention sessions i.e. planning to move, transportation issues
* Neurological disorder pre- or post- stroke affecting subject's ability to follow study directions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lin, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (1):
- Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin C, Morgan CJ, Fortenberry ELS, Androulakis XM, McGregor K. The safety and feasibility of a pilot randomized clinical trial using combined exercise and neurostimulation for post-stroke pain: the EXERT-Stroke study. Front Neurol. 2025 Apr 24;16:1524004. doi: 10.3389/fneur.2025.1524004. eCollection 2025. PMID 40343185

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS+Exercise | Sham rTMS+Exercise
Started | 5 | 4
Completed | 4 | 2
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS+Exercise | Sham rTMS+Exercise | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.9) | 59.9 (7.6) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 3 | 1 | 4
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rankin Scale From Baseline to Follow-up 30 Days After Last Intervention
Description: The modified Ranking scale (mRS) is a single-item, global, Likert-type scale ranging from 0-6 (higher scores mean a worse outcome) to categorize level of functional independence with comparison to pre-stroke function, accounting for activities of daily living. Participants were scored at baseline and 30 days after last intervention.
Time Frame: From baseline to follow-up 30 days after last intervention
Population: Only participants completing both the baseline and followup mRS assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active rTMS+Exercise: Patients with post-stroke headaches.
  Active arm: active rTMS and exercise
- Sham rTMS+Exercise: Patients with post-stroke headaches.
  Control arm: Sham rTMS and exercise arm.
Arm/Group | Active rTMS+Exercise | Sham rTMS+Exercise
Number analyzed (Participants) | 4 | 2
units on a scale | 0 (0) | 1 (1.41)
Statistical Analysis 1: Comparison: Active rTMS+Exercise vs Sham rTMS+Exercise; Test type: Superiority; p = 0.896, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: During the 10 intervention sessions over a 30-day period and a 1-month post-intervention follow-up.
Arm/Group | Active rTMS+Exercise | Sham rTMS+Exercise
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT04672044/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT04672044/ICF_000.pdf